CLINICAL TRIAL: NCT00303992
Title: Weekly Trastuzumab (Herceptin) and Irinotecan in Patients With HER-2 Positive Advanced Breast Cancer: A Phase II Trial
Brief Title: Trastuzumab and Irinotecan in Treating Patients With HER2/Neu Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 037517; UCSF-037517; UCSF-H6961-24269-02A; NCT00145821 (obsolete NCT alias)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trastuzumab and Irinotecan (Experimental)
  Interventions: Biological: trastuzumab; Drug: irinotecan hydrochloride

INTERVENTIONS:
Biological: trastuzumab
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving trastuzumab together with irinotecan may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving trastuzumab together with irinotecan works in treating patients with HER2/neu positive metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall objective response-rate (partial and complete) and stable disease rate in patients with HER2/neu positive metastatic breast cancer treated with the combination of irinotecan hydrochloride and trastuzumab (Herceptin®) after prior first- or second-line therapy with trastuzumab combined with other chemotherapeutic agents.

Secondary

* Determine the toxicities of this combination regimen.
* Determine the duration of response and time to disease progression in patients treated with this combination.
* Document development of brain metastases or progression of known metastases in patients treated with this regimen.

OUTLINE: Patients receive trastuzumab (Herceptin®) IV over 30-90 minutes on days 1, 8, 15, and 22 and irinotecan hydrochloride IV over 30-60 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic breast carcinoma
* Received 1-3 prior chemotherapy regimens for metastatic disease

  * Documented progressive disease
  * Repeated courses of the same chemotherapy agent alone or in combination are considered a single regimen
  * Prior trastuzumab (Herceptin®) alone or with chemotherapy allowed

    * Other biologic agents are not considered a chemotherapy regimen
* Measurable disease

  * Patients with bone-only disease who are evaluable by tumor markers (e.g., CA15-3, CEA, or CA27.29) are eligible

    * Patients must have prior evidence of correlation of disease activity with changes in tumor marker level
* Confirmation of HER2/neu status by a positive test for gene amplification by fluorescence in situ hybridization or 3+ by immunohistochemistry
* Brain metastases allowed if the following criteria are met:

  * Brain metastases were previously treated and are currently stable as documented by head CT scan with contrast or MRI within 4 weeks of study entry

    * Patients with existing brain metastases should have stability documented by prior imaging ≥ 8 weeks before the baseline scan
* Hormone-receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status ≤ 2
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Life expectancy ≥ 12 weeks
* No history of congestive heart failure
* Documented ejection fraction ≥ 45% by MUGA scan or echocardiogram within 1 month of study entry
* Total bilirubin < 3 times upper limit of normal (ULN)
* AST < 3 times ULN (5 times ULN if due to liver involvement)
* Creatinine < 1.5 times ULN
* No history of serious adverse events related to trastuzumab
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No severe, concurrent illness that would prevent compliance with study protocol
* No chronic severe diarrheal illness
* No history of Gilbert's disease or known deficiency in glucuronidation
* No recent or current history of alcoholism or acute viral hepatitis

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No chemotherapy or hormonal therapy within the past 2 weeks
* Prior or concurrent bisphosphonates allowed
* No prior irinotecan (other camptothecins allowed)
* No concurrent radiotherapy
* No ongoing treatment with any other investigational agent

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-05; Primary Completion 2006-11-16 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Overall objective response rate (partial and complete responses) | up to 20 months post treatment
Stable disease rate | up to 20 months post treatment

SECONDARY OUTCOMES:
Toxicity | up to 20 months post treatment
Duration of response | up to 20 months post treatment
Time to disease progression | up to 20 months post treatment
Development of brain metastases or progression of known metastases on this treatment | up to 20 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hope S. Rugo, MD, Principal Investigator — University of California, San Francisco; Judy M. Cheng, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States